CLINICAL TRIAL: NCT06834412
Title: [68Ga]Pentixafor PET/CT for Staging of Hematological Malignancies: Comparison to [18F]FDG PET/CT
Brief Title: A Study Evaluating the Value of 68Ga-Pentixafor PET Imaging in the Staging of Hematological Tumor, and Comparing It with 18F-FDG PET/CT Imaging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: KY20212119-F-1; KY20212119-F-1 (Other: medical ethics committee of the Xijing hospital)
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-09

CONDITIONS: Hematological Malignancies
Keywords: 68Ga-Pentixafor; hematological malignancies; 18F-FDG; staging
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: before-after study in the same patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- before-after study in the same patient (Experimental): This is a prospective, open-label, single-center clinical study for hematological malignancies. 120 patients confirmed by pathology of having NHLs or myeloma were included. Qualified subjects underwent 18F-FDG and 68Ga-Pentixafor PET/CT scans within 7 days after recruited. Patient medical history was collected and laboratory tests were performed before the examination, and a biopsy or surgery was performed to obtain pathological results within 1 month after the examination, followed by a 6-month follow-up. The pathological results were used as the diagnostic gold standard.
  Interventions: Diagnostic Test: 68Ga-Pentixafor and 18F-FDG PET/CT Scan

INTERVENTIONS:
Diagnostic Test: 68Ga-Pentixafor and 18F-FDG PET/CT Scan — The imaging agent 68Ga-Pentixafor and 18F-FDG used in this project is synthesized following the standards for radiopharmaceutical production, with reference to the Chinese Pharmacopoeia (quality standards for 18F-FDG). The pH value is about 4; the radiochemical purity is not less than 95%, and the bacterial endotoxin content in each milliliter of solution is less than 15EU; the radioactive concentration is not less than 37 MBq/mL; the solvent residues comply with the regulations. Specification: 185~1850 MBq/ml Characteristics: Clear, colorless, no visible particles. Radioactive physical half-life: 68Ga is 68 minutes. Expiry: Calculated from the time of labeling, stable for 3 half-lives. Administration method: Intravenous injection. Dosage: 0.05-0.1mCi/kg, flush with 5 mL of saline after injection.

SUMMARY:
This is a prospective, open-label, single-center clinical study targeting hematological malignancies. 120 patients with a confirmed by pathology of non-Hodgkin's lymphoma or myeloma were included. Qualified subjects will undergo 18F-FDG PET/CT and 68Ga-Pentixafor PET/CT examination. The aim is to To investigate whether 68Ga-pentixafor PET imaging can be used as a reliable complement to 18F-FDG PET imaging for clinical staging, treatment response evaluation, and re-staging of patients with hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

Ages 18 to 75 years old Confirmed by pathology with NHLs or myeloma Willing and able to follow the study protocol.

Exclusion Criteria:

Children, pregnant or lactating women Severely impaired liver and kidney function (alanine aminotransferase > 8-10 times the upper limit of normal, serum creatinine 186-442 umol/L) With a history of allergy to contrast media or other drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Standardized uptake value (SUVmax) | 1 day from injection of the tracer
  Maximum Standardized uptake value (SUVmax) of [68Ga]Pentixafor and [18F]FDG in the included subjects' primary and/or metastatic lesions.
Mean Standardized Uptake Value(SUVmean) of liver | 1 day from injection of the tracer
  Mean Standardized uptake value (SUVmean) of [68Ga]RCCB6 and [68Ga]PSMA in the included subjects' liver.
Mean Standardized uptake value (SUVmean) | 1 day from injection of the tracer
  Mean Standardized uptake value (SUVmean) of [68Ga]Pentixafor and [18F]FDG in the included subjects' primary and/or metastatic lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- Department ofNuclear Medicine,Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu X, Tang H, Ou H, Quan Z, Li G, Gao G, Wang J, Kang F. Establishment and validation of a clinical threshold criteria for choosing PET imaging tracers for indolent non-Hodgkin's lymphoma. EJNMMI Res. 2025 Dec 27. doi: 10.1186/s13550-025-01368-7. Online ahead of print. PMID 41455028